CLINICAL TRIAL: NCT06198101
Title: Effects of Myofascial Release Technique With and Without Segmental Vibrator on Upper Limb Functions in Children With Spastic Cerebral Palsy
Brief Title: Effects of Myofascial Release Technique on Upper Limb Functions in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0745
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: CP child; Myofascial release technique; Segmental vibrator
MeSH Terms: conditions — Cerebral Palsy | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: It will be Randomized control trial in which non probabilty convenient sampling will be used. Two groups of 6-12 age will be formed in which participants will be randomly divided. Group A will only receive Myofascial release technique and group B will receive Myofascial release technique with segmental massage vibrator
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial release technique (Active Comparator): This group receive Myofascial Release Technique
  Interventions: Other: Myofascial Release Technique
- Myofascial Release Technique along with segmental massage vibrator (Experimental): this group receive Myofascial Release Technique along with segmental massage vibrator
  Interventions: Other: Myofascial Release Technique along with segmental vibrator

INTERVENTIONS:
Other: Myofascial Release Technique — The treatment will be applied by the therapist standing at the side of the patient with different levels according to subject's tolerance for duration of 3 minutes in each sitting. Level one will be performed by longitudinal movements without causing any tension to the tissues. The level two will be performed by longitudinal movements with light pressure to the tensed muscle. The level three will be performed by compressing the treatment area then passively fullest possible range of motion will be performed and then longitudinal movement will be done with same compression. In level four, the patient will actively move the tissue through the fullest possible range of motion. The taut band will palpate and then firm pressure will be maintained and then longitudinal movements will be performed. Treatment will be applied for two intervention sessions per week and a total of 12 sessions over 6 weeks.
  Arms: myofascial release technique
Other: Myofascial Release Technique along with segmental vibrator — this group will receive vibratory stimulations through segmental vibrator along the muscle fibers of upper limb flexors, extensors, and wrist flexors for 10-minutes each session with low amplitude (0.3-0.5 mm peak to peak) at fixed frequency of 150 Hz(23). Along with segmental vibrator group B will also receive myofascial release technique through the same method to the upper limb flexors, extensors, and wrist flexors. Group B will receive both treatments for two intervention sessions per week and a total of 12 sessions over 6 weeks.
  Arms: Myofascial Release Technique along with segmental massage vibrator

SUMMARY:
Cerebral palsy (CP) is a common neurodevelopmental disorder characterized by motor impairments, including spasticity, muscle tightness, and limited range of motion in the limbs. Myofascial Release Technique (MRT) has shown promise as a non-invasive intervention for addressing musculoskeletal dysfunctions and improving range of motion in various populations.

The study will employ a randomized controlled trial design to investigate the effects of myofascial release technique (MRT) with and without a segmental vibrator on upper limb functions in children with spastic cerebral palsy (CP). The study will be conducted at PSRD and Rising Sun Institute Lahore. A sample of children aged 6-12 years with a diagnosis of spastic CP will be recruited and randomly assigned to two groups: MRT with a segmental vibrator, and MRT without a segmental vibrator. The MRT interventions will be provided by trained therapists for a specified duration and frequency over a period of 4 weeks. Spasticity will be measured by the Modified Ashwarth Scale, Upper limb extremity function via Pediatric Upper Extremity Motor Activity Log-Revised (PMAL), and range of motion will be assessed by Goniometer. Data will be analyzed using appropriate statistical tests to determine the effects of the interventions on upper limb functions in children with spastic CP. Ethical considerations will be followed, and informed consent will be obtained from the participant's parents or legal guardians.

DETAILED DESCRIPTION:
Group A will receive only myofascial release technique through longitudinal sliding and cross handed held method to the upper limb flexors, extensors, and wrist flexors. The treatment will be applied by the therapist standing at the side of the patient. Then technique will be applied with different levels according to subject's tolerance for duration of 3 minutes in each sitting. Level one will be performed by longitudinal movements without causing any tension to the tissues. The level two will be performed by longitudinal movements with light pressure to the tensed muscle. The level three will be performed by compressing the treatment area then passively fullest possible range of motion will be performed and then longitudinal movement will be done with same compression. In level four, the patient will actively move the tissue through the fullest possible range of motion. The taut band will palpate and then firm pressure will be maintained and then longitudinal movements will be performed. Treatment will be applied for two intervention sessions per week and a total of 12 sessions over 6 weeks.

Group B will receive vibratory stimulations through segmental vibrator along the muscle fibers of upper limb flexors, extensors, and wrist flexors for 10-minutes each session with low amplitude (0.3-0.5 mm peak to peak) at fixed frequency of 150 Hz. Along with segmental vibrator group B will also receive myofascial release technique through the same method to the upper limb flexors, extensors, and wrist flexors. Group B will receive both treatments for two intervention sessions per week and a total of 12 sessions over 6 weeks.

ELIGIBILITY:
Inclusion Criteria

* Children aged 6-12 years.
* Both Boys and Girls
* Spasticity above 1+ grade of ashworth scale
* Ability to follow instructions and participate in therapy sessions

Exclusion Criteria:

* Unable to follow command.
* Multiple Musculoskeletal deformities or contractures that may limit upper limb function.
* Children who are Contraindicated to myofascial release technique or the use of a segmental vibrator for example burn.
* Recent upper limb surgery or significant upper limb injuries.
* Participation in any other concurrent therapy or intervention for upper limb function.
* Inability to commit to the study protocol or attend scheduled therapy sessions

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Modified Ashwarth Scale | 6 weeks
  The Modified Ashworth Scale (MAS) is a commonly used clinical assessment tool to evaluate muscle tone and spasticity in individuals with neurological conditions such as spastic cerebral palsy. It is a reliable and valid method for grading muscle resistance during passive movement(18). interrater reliability of AS and MAS varied from moderate to good. ICC scores of AS were between 0.54 and 0.78 and MAS were between 0.61-0.87. Test-retest results of AS and MAS varied from poor to good. ICC values were between 0.31 and 0.82 for AS and between 0.36 and 0.83 for MAS
The Pediatric Upper Extremity Motor Activity Log-Revised (PMAL) | 6 weeks
  this tool is a validated assessment tool designed to measure the quality and quantity of upper extremity use in children with neurological conditions, including spastic cerebral palsy(19). The PMAL consists of a structured interview and a 28-item questionnaire that assesses how frequently and how well a child uses their upper limb in various daily activities. The PMAL has demonstrated good reliability (n=0.91) and validity (r= 05) and has been widely used in research and clinical practice to evaluate upper extremity function and monitor progress in rehabilitation interventions. It offers valuable insights into the effectiveness of therapeutic interventions and helps guide treatment planning and goal setting for children with spastic CP
Goniometer | 6 weeks
  : A goniometer is a measurement tool commonly used in rehabilitation and physical therapy to assess the range of motion (ROM) of various joints in the body. It consists of a stationary arm and a movable arm with a protractor-like scale, allowing for precise measurement of joint angles. By aligning the stationary arm with the joint's axis and the movable arm with the body segment, the goniometer provides objective measurements of joint flexibility, mobility, and muscle strength. The goniometer provides valuable quantitative data that can guide treatment planning, monitor patient progress, and assess functional outcomes related to joint movement and mobility

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Mangrio, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah JP, Thaker N, Heimur J, Aredo JV, Sikdar S, Gerber L. Myofascial Trigger Points Then and Now: A Historical and Scientific Perspective. PM R. 2015 Jul;7(7):746-761. doi: 10.1016/j.pmrj.2015.01.024. Epub 2015 Feb 24. PMID 25724849